CLINICAL TRIAL: NCT02286115
Title: Life-Stress Interview for Women With Chronic Urogenital Pain Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC.2014-151
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Urogenital Pain
Keywords: Chronic Pelvic Pain; Interstitial Cystitis; Vulvodynia; Dyspareunia; Pelvic Floor Dysfunction; Emotional Processing
MeSH Terms: conditions — Cystitis, Interstitial; Vulvodynia; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Life-Stress Interview (Experimental): The Life-Stress Interview is an experiential assessment technique
  Interventions: Behavioral: Life-Stress Interview
- Wait-list Control (No Intervention): Wait-list Control

INTERVENTIONS:
Behavioral: Life-Stress Interview — A life-stress interview which aims to help patients: a) disclose their stressful experiences and emotional conflicts, which might be contributing to their symptoms, b) learn about associations between their stress and physical symptoms; and c) learn about the potential value of experiencing and expressing their emotions related to these stressful situations
  Arms: Life-Stress Interview

SUMMARY:
The goal of this study is to test the efficacy, feasibility, and acceptability of providing an experiential assessment interview that targets health, and emotional and stressful experiences in a tertiary care setting specializing in women's urology.

DETAILED DESCRIPTION:
In this randomized, controlled trial, the investigators will compare an interview condition to a wait-list control condition. The investigators hypothesize that helping individuals identify the links between their stress, emotions, and physical symptoms will likely increase their awareness and endorsement of the link between stress and physical symptoms, including a willingness to engage in stress management techniques. It is also expected that helping raise an individual's awareness about their symptoms, followed by an experience and expression of unexpressed emotion is likely to influence their physical and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a chronic urogenital pain condition

Exclusion Criteria:

* non-English speaking
* unable to read
* psychosis
* dementia
* mental impairment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Symptom Interpretation Questionnaire (SIQ) | Change from baseline symptom attribution at 6-weeks
Brief Pain Inventory (BPI) | Change from baseline pain at 6-weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire-15 (PHQ-15) | Change from baseline in symptom severity at 6 weeks
Brief Symptom Inventory (BSI) | Change from baseline symptoms at 6-weeks
Satisfaction With Life Scale (SWLS) | Change from baseline life satisfaction at 6-weeks
Pelvic Floor Distress Inventory -20 (PFDI-20) | Change from baseline pelvic symptoms at 6-weeks
Global Assessment Response (GRA) | Change from baseline overall symptoms at 6-weeks
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) | Change from baseline pain at 6-weeks
Emotional Approach Coping (EAC) | Change from baseline emotional approach coping at 6-weeks
Emotional Processing Scale-25 (EPS-25) | Change from baseline emotional processing at 6-weeks
Inventory of Interpersonal Problems-32 (IIP-32) | Change from baseline interpersonal problems at 6-weeks
Pain Catastrophizing Scale | Change from baseline pain catastrophizing at 6-weeks
Change Assessment Questionnaire | Change from baseline stage of change at 6-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Carty, M.A., Principal Investigator — Beaumont Health Systems and Wayne State University; Mark A Lumley, PhD, Principal Investigator — Wayne State University
Locations (1):
- Women's Urology Center, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597